CLINICAL TRIAL: NCT01832636
Title: Intervention and Mechanisms of Alanyl-Glutamine for Inflammation, Nutrition, and Enteropathy (IMAGINE)
Brief Title: Intervention and Mechanisms of Alanyl-Glutamine for Inflammation, Nutrition, and Enteropathy
Acronym: IMAGINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Universidade Federal do Ceara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN001 -"IMAGINE"
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Malnutrition; Environmental Enteropathy; Diarrhea
Keywords: L-Alanyl-L-Glutamine; Environmental enteric dysfunction; Tropical enteropathy
MeSH Terms: conditions — Malnutrition; Diarrhea; Sprue, Tropical | interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Alanyl-Glutamine 3g/d (Active Comparator): Alanyl-Glutamine orally 3g/day for 10 days
  Interventions: Dietary Supplement: Alanyl-Glutamine
- Alanyl-Glutamine 6g/d (Active Comparator): Alanyl-Glutamine orally 6g/day for 10 days
  Interventions: Dietary Supplement: Alanyl-Glutamine
- Alanyl-Glutamine 12g/d (Active Comparator): Alanyl-Glutamine orally 12g/d for 10 days
  Interventions: Dietary Supplement: Alanyl-Glutamine
- Glycine 12.5g/d (Placebo Comparator): Glycine orally 12.5 g/d for 10 days. This dose is calculated to be isonitrogenous to 12g of Alanyl-Glutamine.
  Interventions: Dietary Supplement: Alanyl-Glutamine

INTERVENTIONS:
Dietary Supplement: Alanyl-Glutamine — Alanyl-Glutamine and Glycine doses will be prepared immediately prior to administration by dissolving in formula, milk, or fruit juice. Administration of each dose will be directly observed by a study nurse or health agent.
  Other Names: AminoStable (Ajinomoto)

SUMMARY:
Several host factors underlie the pathogenesis of the reciprocal cycle of childhood diarrhea and undernutrition in developing countries. These include intestinal inflammation, mucosal damage, and alterations in intestinal barrier function that lead to malabsorption, growth failure, and heightened susceptibility to recurrent and prolonged episodes of diarrhea. Recent studies from Northeast Brazil demonstrate the benefits of a novel alanyl-glutamine-based oral rehydration and nutrition therapy (Ala-Gln ORNT) in speeding the recovery of damaged intestinal barrier function in cell culture, animal models, patients with AIDS, and underweight children.

Oral supplementation with Alanyl-Glutamine (Ala-Gln; 24g a day for 10 days) improves short-term gut integrity and weight velocity 4 months after therapy in a group of undernourished children from Northeast Brazil. Intervention and Mechanisms of Alanyl-Glutamine for Inflammation, Nutrition, and Enteropathy (IMAGINE) is a study designed to answer the following questions: 1) What is the lowest dose of Ala-Gln that improves intestinal barrier function, intestinal inflammation, and nutritional status in children at risk of underweight, wasting, or stunting? 2) What are the mechanisms by which Ala-Gln exerts these benefits?

ELIGIBILITY:
Inclusion Criteria:

1. Children who are undernourished or at risk of undernutrition, with anthropometric z-scores less than or equal to -1 for one of these parameters: height-for-age, weight-for-age, or weight-for-height.
2. Children ages 2 months to 5 years old.

Exclusion Criteria:

1. Children who are exclusively breastfed.
2. Have participated in another intervention study in the past two years.
3. Fever greater than 38.8 ° C.
4. Use of antibiotics.
5. Systemic disease or other serious medical condition (including, but not limited to meningitis, pneumonia, tuberculosis, and chickenpox).
6. Children who are unable to ingest, retain or absorb nutritional supplements.
7. Children whose families plan to move from the study area within the next 6 months.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Urinary Lactulose: Mannitol Intestinal Permeability Test | Urine Collection on Day 1, 10-13, 30-37
  Determine the dose-and time-effect of alanyl-glutamine on intestinal barrier function recovery using the intestinal permeability test, with measurement of the percentage of urinary excretion of lactulose, mannitol and ratio of lactulose:mannitol.

SECONDARY OUTCOMES:
Fecal Lactoferrin Test | Fecal sample collected on Day 1, 10-13, 30-37
  To evaluate the effect of time and dose-response of alanyl-glutamine on intestinal inflammation, as measured by qualitative or quantitative testing for fecal lactoferrin in stools of children at risk of undernutrition.
Fecal Cytokine Measurement | Fecal sample collected on Day 1, 10-13
  To evaluate the effect of alanyl-glutamine on intestinal inflammation, by measuring proinflammatory cytokines interleukin-1, interleukin-8, tumor necrosis factor-alpha (TNF), and regenerating gene 1B (REG1B) in stools of children at risk of undernutrition.
Anthropometry | Measured and calculated Day 1, 10-13, 30-37, 90-104, 120-141
  To evaluate the time and dose-effect of alanyl-glutamine on short and medium-term nutritional status by evaluating changes in anthropometric measures (z scores) over time: height-for-age, weight-for-age, and weight-for-height.
Fecal Calorimetry | Fecal sample collected on Day 1, 10-13, 30-37
  To evaluate the effect of time and dose-response of alanyl-glutamine on the intestinal absorption of fat, protein, and carbohydrates, by measurement of fecal energy content by bomb calorimetry.
Metabolomic Profile of Urine | Collected on Day 1, 10-13, 30-37
  To evaluate the time and dose-effect of alanyl-glutamine on metabolism in children at risk of undernutrition by means of urine metabolomic profile tests.
History of Diarrhea in the Previous Two Weeks | Day 1, 30-37, 90-104, 120-141
  History of diarrhea in the previous two weeks. A day of diarrhea will be defined as 3 or more looser than normal bowel movements in a 24-hour period. Distinct episodes must be separated by at least 2 days without diarrhea. Duration of episodes will be classified as acute (< 7 days), prolonged acute (>6 and <14 days), or persistent (>13 days).

CONTACTS AND LOCATIONS:
Overall Officials: Sean R Moore, MD, MS, Principal Investigator — Cincinnati Children´s Hospital; Aldo Lima, MD, PhD, Principal Investigator — Universidade Federal do Ceara
Locations (1):
- Universidade Federal do Ceara, Fortaleza, Ceará, Brazil

REFERENCES:
- [Background] Lima NL, Soares AM, Mota RM, Monteiro HS, Guerrant RL, Lima AA. Wasting and intestinal barrier function in children taking alanyl-glutamine-supplemented enteral formula. J Pediatr Gastroenterol Nutr. 2007 Mar;44(3):365-74. doi: 10.1097/MPG.0b013e31802eecdd. PMID 17325559
- [Derived] Moore SR, Quinn LA, Maier EA, Guedes MM, Quetz JS, Perry M, Ramprasad C, Lanzarini Lopes GML, Mayneris-Perxachs J, Swann J, Soares AM, Filho JQ, Junior FS, Havt A, Lima NL, Guerrant RL, Lima AAM. Intervention and Mechanisms of Alanyl-glutamine for Inflammation, Nutrition, and Enteropathy: A Randomized Controlled Trial. J Pediatr Gastroenterol Nutr. 2020 Sep;71(3):393-400. doi: 10.1097/MPG.0000000000002834. PMID 32826717